CLINICAL TRIAL: NCT05310916
Title: Evaluation of the Effect of Sodium-Glucose Cotransporter-2 (SGLT2) Inhibitors on Diabetic Retinopathy in Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of SGLT2i on Diabetic Retinopathy in Type 2 Diabetes Mellitus Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nidae Alaa (Other)
Responsible Party: Sponsor-Investigator, Nidae Alaa, Principal Investigator, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 311311
Record Dates: First submitted 2022-03-27; First posted 2022-04-05 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic retinopathy; Sodium-glucose cotransporter-2 inhibitor
MeSH Terms: conditions — Diabetic Retinopathy | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): (n=30): type 2 diabetes mellitus patients who will receive an oral antidiabetic along with dapagliflozin at a dose of 10 mg daily for 12 weeks.
  Interventions: Drug: Dapagliflozin 10mg Tab plus another oral hypoglycemic agent
- Control group (Active Comparator): (n=30): type 2 diabetes mellitus patients who will receive two oral antidiabetic agents for 12 weeks
  Interventions: Drug: Two oral hypoglycemic agents other than dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab plus another oral hypoglycemic agent — Dapagliflozin is a member of Sodium-glucose co-transporter 2 inhibitors class which in addition to its glucose control effect, has reno-protective and cardioprotective effects, controls blood pressure and causes weight loss.
  Other Names: Diglifloz 10mg Tab
  Arms: Test group
Drug: Two oral hypoglycemic agents other than dapagliflozin — Two oral anti-diabetic agents not including sodium-glucose co-transporter 2 inhibitors
  Other Names: Oral anti-diabetic agents
  Arms: Control group

SUMMARY:
A prospective, randomized, open-label, controlled clinical trial will be conducted at the endocrinology department - Ain Shams University (ASU) hospital. Sixty patients will be enrolled into the study. 30 of which will receive dapagliflozin 10mg tab once daily and the other thirty will receive their standard antidiabetic therapy for 12 weeks.

DETAILED DESCRIPTION:
All type 2 diabetes mellitus patients presenting to the endocrinology department, ASU Hospitals, who were diagnosed with mild to moderate non-proliferative diabetic retinopathy will be assessed for eligibility.

Eligible patients will be randomly assigned to one of the following 2 arms:

1. Group 1 (Control group) (n= 30): type 2 diabetes mellitus patients who will receive their oral antidiabetic for 12 weeks.
2. Group 2 (Test group) (n= 30): type 2 diabetes mellitus patients who will receive their oral antidiabetic along with dapagliflozin at a dose of 10 mg daily for 12 weeks.

A total of four visits one for baseline evaluation and one for end of study evaluation and two intermediate visits, the following will be performed in the visits:

1. Clinical Evaluation

   1. Systolic and diastolic blood pressures recording.
   2. Plasma glucose measurement.
2. Report any adverse effects that may appear
3. Blood samples will be taken at baseline and at 12-week visits
4. Follow up

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged between 40 and 70 years old.
2. Glomerular filtration rates > 60 mL/min.
3. Normal aspartate and alanine transaminase levels.
4. Controlled systolic and diastolic blood pressures

Exclusion Criteria:

1. Patients using insulin or more than one oral anti-diabetic drug.
2. Patients who have HbA1c level ≥10% (86 mmol/mol) or a fasting plasma glucose level >240 mg/dl.
3. Patients with a history of cardiovascular events within six months before enrolment.
4. Patients suffering from cataract or glaucoma.
5. Patients with volume depletion clinical signs.
6. Body mass index (BMI) >40 kg/m2
7. Infectious or inflammatory diseases.
8. Neoplasm, or hematological disorders.
9. Pregnant or breast-feeding patients.
10. Active participation in another clinical study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Severity of retinopathy | 12 weeks
  evaluate the change of stage of disease according to diabetic retinopathy severity scale,, Which is the International Clinical Disease Severity Scale (ICDSS) for DR. This scale classified the severity of disease into five stages ( No apparent retinopathy, Mild Non proliferative Diabetic retinopathy (NPDR) ,Mod NPDR, Severe NPDR ,Proliferative Diabetic Retinopathy) depend on eye examination. higher scores mean worse outcome.
Evaluation of the study biomarkers, IL-6, and VEGF | 12 weeks
  Interleukin-6 (IL-6)//inflammatory biomarker Vascular endothelial growth factor (VEGF)//angiogenic biomarker

SECONDARY OUTCOMES:
Occurrence of adverse events | (1-90)days
  No potential risks are expected when the study patients are selected according to the determined inclusion criteria but maybe occur Nausea, abdominal pain, polyuria, thrush, genital or urinary tract infections

CONTACTS AND LOCATIONS:
Overall Officials: Lamiaa M ElWakeel, PhD, Study Director — Faculty of pharmacy Ain Shams University; Mona A Abd El Salam, MD, Study Director — Faculty of Medicine Ain Shams University; Marwa A Ahmed, PhD, Study Director — Faculty of pharmacy Ain Shams University; Nidae A Ismail, BSc, Principal Investigator — Faculty of pharmacy Ain Shams University
Locations (1):
- Internal medicine and endocrinology department, Ain-shams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zheng Y, Ley SH, Hu FB. Global aetiology and epidemiology of type 2 diabetes mellitus and its complications. Nat Rev Endocrinol. 2018 Feb;14(2):88-98. doi: 10.1038/nrendo.2017.151. Epub 2017 Dec 8. PMID 29219149
- [Background] Wong TY, Cheung CM, Larsen M, Sharma S, Simo R. Diabetic retinopathy. Nat Rev Dis Primers. 2016 Mar 17;2:16012. doi: 10.1038/nrdp.2016.12. PMID 27159554
- [Background] Sha W, Wen S, Chen L, Xu B, Lei T, Zhou L. The Role of SGLT2 Inhibitor on the Treatment of Diabetic Retinopathy. J Diabetes Res. 2020 Nov 12;2020:8867875. doi: 10.1155/2020/8867875. eCollection 2020. PMID 33274239
- [Background] Zhou Z, Ju H, Sun M, Chen H. Serum Vascular Endothelial Growth Factor Levels Correlate with Severity of Retinopathy in Diabetic Patients: A Systematic Review and Meta-Analysis. Dis Markers. 2019 Mar 24;2019:9401628. doi: 10.1155/2019/9401628. eCollection 2019. PMID 31019585
- [Background] Yao Y, Li R, Du J, Long L, Li X, Luo N. Interleukin-6 and Diabetic Retinopathy: A Systematic Review and Meta-Analysis. Curr Eye Res. 2019 May;44(5):564-574. doi: 10.1080/02713683.2019.1570274. Epub 2019 Feb 4. PMID 30644770
- [Background] Peters AL, Buschur EO, Buse JB, Cohan P, Diner JC, Hirsch IB. Euglycemic Diabetic Ketoacidosis: A Potential Complication of Treatment With Sodium-Glucose Cotransporter 2 Inhibition. Diabetes Care. 2015 Sep;38(9):1687-93. doi: 10.2337/dc15-0843. Epub 2015 Jun 15. PMID 26078479
- [Background] Lahoti S, Nashawi M, Sheikh O, Massop D, Mir M, Chilton R. Sodium-glucose co-transporter 2 inhibitors and diabetic retinopathy: insights into preservation of sight and looking beyond. Cardiovasc Endocrinol Metab. 2020 May 18;10(1):3-13. doi: 10.1097/XCE.0000000000000209. eCollection 2021 Mar. PMID 33634250
- [Background] Chen YY, Wu TT, Ho CY, Yeh TC, Sun GC, Kung YH, Wong TY, Tseng CJ, Cheng PW. Dapagliflozin Prevents NOX- and SGLT2-Dependent Oxidative Stress in Lens Cells Exposed to Fructose-Induced Diabetes Mellitus. Int J Mol Sci. 2019 Sep 5;20(18):4357. doi: 10.3390/ijms20184357. PMID 31491943
- [Background] Ott C, Jumar A, Striepe K, Friedrich S, Karg MV, Bramlage P, Schmieder RE. A randomised study of the impact of the SGLT2 inhibitor dapagliflozin on microvascular and macrovascular circulation. Cardiovasc Diabetol. 2017 Feb 23;16(1):26. doi: 10.1186/s12933-017-0510-1. PMID 28231831
- See also: Protective Effect of Sodium-Glucose Co-Transporter 2 Inhibitor (Dapagliflozin) on Diabetic Retinopathy in Streptozotocin Induced Diabetes in Rats — https://mjcu.journals.ekb.eg/article_52382.html